CLINICAL TRIAL: NCT07324499
Title: Effect of Dexamethasone on Plasma Levels of Bupivacaine and Dexamethasone Following a Single-injection Interscalene Nerve Block: A Randomized Controlled Study
Brief Title: Effect of Dexamethasone on Plasma Levels of Bupivacaine and Dexamethasone After a Single-injection Interscalene Nerve Block.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 250429018
Record Dates: First submitted 2025-12-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Pain; Interscalene Blocks; Dexamethasone; Bupivacaine
Keywords: Dexamethasone; Bupivacaine; Pain; Interscalene blocks
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous dexamethasone (Active Comparator): cccc
  Interventions: Drug: administration of dexamethasone intravenously
- Local dexamethasone (No Intervention): ccc

INTERVENTIONS:
Drug: administration of dexamethasone intravenously — IV dexamethasone administration will be added to the interscalene block. In the control group, dexamethasone will be applied perineurally.
  Arms: Intravenous dexamethasone

SUMMARY:
Recent studies have highlighted the comparative advantages of perineural dexamethasone, particularly regarding its safety profile and its ability to prolong analgesia in various peripheral nerve blocks. A recent systematic review demonstrated that perineural administration of dexamethasone significantly extends the duration of analgesia compared to intravenous administration.

The mechanism of action of perineural dexamethasone remains unclear. Moreover, there is a lack of research comparing the systemic absorption of local anesthetics administered perineurally with or without dexamethasone, and the systemic absorption and bioavailability of dexamethasone when used as a perineural adjuvant have not been studied.

Objective: This study aims to compare plasma concentrations of bupivacaine following a single-shot interscalene block with dexamethasone administered either perineurally or intravenously.

Methodology: A prospective, randomized, double-blind trial will be conducted involving 40 patients undergoing shoulder surgery requiring a single-shot interscalene block. Each patient will receive 20 mL of 0.25% bupivacaine combined with 8 mg of dexamethasone administered either perineurally or intravenously. Venous blood samples (5 mL) will be collected at 5, 10, 20, 40, 80, 120, and 240 minutes post-block, and one sample at discharge, to measure plasma concentrations of both enantiomers of bupivacaine (D(+)-bupivacaine and L(-)-bupivacaine) and dexamethasone.

Outcomes: The study will compare plasma levels of bupivacaine between groups, characterize the pharmacokinetics of bupivacaine and dexamethasone, and assess block duration and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

- ASA I-II patients, with a body mass index (BMI) between 20 and 34 kg/m2 scheduled for shoulder surgery requiring single-needle interscalene block

Exclusion Criteria:

- Chronic opioid use, liver failure, kidney failure, allergy to protocol drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
plasma levels of bupivacaine between groups | 4 hours
  Plasma levels of bupivacaine after a single-shot interscalene block combined with dexamethasone administration ev or perineurally